CLINICAL TRIAL: NCT01761786
Title: Cost-effectiveness of CYP2C19 Genotype Guided Treatment With Antiplatelet Drugs in Patients With ST-segment-elevation Myocardial Infarction Undergoing Immediate PCI With Stent Implantation: Optimization of Treatment (POPular Genetics).
Brief Title: Cost-effectiveness of Genotype Guided Treatment With Antiplatelet Drugs in STEMI Patients: Optimization of Treatment (POPular Genetics)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vera HM Deneer (Other)
Collaborators: Isala (Other); Meander Medical Center (Other); UMC Utrecht (Other); University Medical Center Groningen (Other); OLVG (Network); Onze Lieve Vrouw Hospital (Other); Amphia Hospital (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Federico II University (Other); Rijnstate Hospital (Other)
Responsible Party: Sponsor-Investigator, Vera HM Deneer, PharmD, PhD, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGxSTEMI08
Record Dates: First submitted 2012-09-19; First posted 2013-01-07 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Myocardial Infarction; STEMI
Keywords: Myocardial Infarction; Thrombosis; Acute Coronary Syndrome; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Embolism and Thrombosis; Genetic Testing; Clopidogrel; Prasugrel; Ticagrelor; Platelet Aggregation Inhibitors; Purinergic P2Y Receptor Antagonists
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Thrombosis; Acute Coronary Syndrome; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Embolism and Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): CYP2C19 genotyping will be performed after end of study. Patients will be treated with prasugrel or ticagrelor, according to local protocol.
- Intervention group (Active Comparator): CYP2C19 genotyping will be performed <48h after PCI and antiplatelet treatment will be chosen based on genotyping results.
  Interventions: Genetic: CYP2C19 genotyping

INTERVENTIONS:
Genetic: CYP2C19 genotyping — CYP2C19 genotyping will be performed in the intervention group. In patients with *1/*1 genotype (Extensive Metabolizer) clopidogrel will be prescribed. All patients who are carrier of a loss-to-function (*2 or *3) gene allel and all patients randomized to the control group will be prescribed prasugrel or ticagrelor, according to local protocol.
  Arms: Intervention group

SUMMARY:
Rationale: the use of antiplatelet drugs (i.e. clopidogrel, ticagrelor or prasugrel) is crucial in the treatment of patients undergoing percutaneous coronary intervention (PCI) with stent implantation to prevent atherothrombotic events. Ticagrelor and prasugrel are more effective in preventing atherothrombotic events, but with a higher risk of bleeding complications, compared to clopidogrel. Clopidogrel is converted into its active metabolite by CYP2C19. Carriers of the non functional CYP2C19*2 and *3 alleles have an impaired CYP2C19 capacity, making clopidogrel less effective. For these subjects ticagrelor or prasugrel is an alternative.

Objective: to assess the efficacy, safety and cost-effectiveness of the CYP2C19 genotype guided antiplatelet treatment strategy, using clopidogrel in non-carriers of a CYP2C19*2 or *3 allele and ticagrelor or prasugrel in carriers of a CYP2C19*2 or *3 allele in STEMI patients.

Intervention: the intervention group will be genotyped for CYP2C19*2 and *3 allele variants within 48 hours after primary PCI. Carriers will receive either ticagrelor (90 mg twice daily) or prasugrel (10 mg once daily or 5 mg once daily if the patient is older than age 75 or has a body weight less than 60 kg), according to local standards. Non-carriers will be treated with clopidogrel (75 mg once daily). The control group receives either ticagrelor or prasugrel, according to local standards at the same dosage as the CYP2C19*2 or *3 carriers in the intervention group. The antiplatelet drug will be continued for one year after PCI. The follow-up duration will be one year using follow-up questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* more than 21 years of age with symptoms of acute myocardial infarction of more than 30 minutes but less than 12 hours
* performed primary PCI with stenting for STEMI

Exclusion Criteria:

* unable to give informed consent or have a life expectancy of less than one year
* active malignancy with increase in bleeding risk, in the investigator's opinion
* women who are known to be pregnant or who have given birth within the past 90 days or who are breastfeeding
* having received thrombolytic therapy within the previous 24 hours or oral anticoagulants during the previous 7 days
* severe renal function impairment needing dialysis
* confirmed or persistent severe hypertension (Systolic Blood Pressure (SBP) > 180 mmHg and/or Diastolic Blood Pressure (DBP) >110 mmHg) at randomization
* contraindication to anticoagulation or at increased bleeding risk, at the investigator's opinion
* cardiogenic shock (SBP ≤ 80mmHg for >30 mins) or Intra-Aortic Balloon Pump (IABP) placed
* history of major surgery, severe trauma, fracture or organ biopsy within 90 days prior to randomisation
* clinically significant out of range values for platelet count or haemoglobin level at screening, in the investigator's opinion.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Net clinical benefit | 1 year
  The primary endpoint is the number of patients who either died, developed a recurrent myocardial infarction (MI), developed definite stent thrombosis, stroke or PLATO major bleeding at 1 year after PCI.
Safety endpoint | 1 year
  The primary safety endpoint is the number of patients with PLATO major or minor bleeding at 1 year after PCI.
Pharmacoeconomics endpoint | 1 year
  The primary endpoints in terms of pharmacoeconomics are quality of life, direct medical costs e.g. costs for blood transfusions, drugs, hospitalization and non-medical costs e.g. costs incurred due to sickness absence.

SECONDARY OUTCOMES:
Net clinical benefit at 30 days | 30 days
  The number of patients who either died, developed a recurrent myocardial infarction (MI), developed definite stent thrombosis, stroke or PLATO major bleeding at 30 days after PCI.
Secondary efficacy and safety endpoint | 30 days and 1 year
  both efficacy and safety will be studied in more detail, using the items of the primary endpoint (death, recurrent myocardial infarction, stentthrombosis, stroke, PLATO major bleeding) as separate parameters and in different combinations, adding cardiovascular and cerebrovascular death, probable and possible stent thrombosis, urgent target vessel revascularization (uTVR) and hospital admission for acute coronary syndrome (ACS) to the efficacy analysis, and (non-)CABG-related bleeding, major-, minor-, life threatening-, fatal-, intracranial and bleeding requiring transfusion to the bleeding analysis, both for 30 days and 1 year follow-up
Secondary safety endpoint | 30 days and 1 year
  Number of patients with bleeding events in 1 year follow up, not only using PLATO bleeding classification, but also, TIMI and BARC bleeding classifications to make the study comparable to previous and future publications
Drug endpoint | 30 days and 1 year
  Comparing the number of patients switching from the recommended P2Y12 inhibitor to a different P2Y12 inhibitor and the number of patients who discontinue the P2Y12 inhibitor early in both the control and genotype group

CONTACTS AND LOCATIONS:
Overall Officials: Jurrien M ten Berg, MD, PhD, FESC, FACC, Principal Investigator — St. Antonius Hospital Nieuwegein, The Netherlands; Daniel MF Claassens, MD, Study Chair — St. Antonius Hospital Nieuwegein, The Netherlands
Locations (10):
- OLV Hospital, Aalst, Belgium
- University of Naples Federico II, Naples, Italy
- Netherlands (8):
  - Meander Medisch Centrum, Amersfoort
  - OLVG, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Amphia Hospital, Breda
  - University Medical Center Groningen, Groningen
  - St. Antonius Hospital, Nieuwegein
  - University Medical Center, Utrecht
  - Isala Klinieken, Zwolle

REFERENCES:
- [Background] Harmsze A, van Werkum JW, Bouman HJ, Ruven HJ, Breet NJ, Ten Berg JM, Hackeng CM, Tjoeng MM, Klungel OH, de Boer A, Deneer VH. Besides CYP2C19*2, the variant allele CYP2C9*3 is associated with higher on-clopidogrel platelet reactivity in patients on dual antiplatelet therapy undergoing elective coronary stent implantation. Pharmacogenet Genomics. 2010 Jan;20(1):18-25. doi: 10.1097/FPC.0b013e328333dafe. PMID 19934793
- [Background] Harmsze AM, van Werkum JW, Ten Berg JM, Zwart B, Bouman HJ, Breet NJ, van 't Hof AW, Ruven HJ, Hackeng CM, Klungel OH, de Boer A, Deneer VH. CYP2C19*2 and CYP2C9*3 alleles are associated with stent thrombosis: a case-control study. Eur Heart J. 2010 Dec;31(24):3046-53. doi: 10.1093/eurheartj/ehq321. Epub 2010 Sep 10. PMID 20833683
- [Background] Peters BJ, Harmsze AM, ten Berg JM, Maitland-van der Zee AH, Tjoeng MM, de Boer A, Deneer VH. CYP2C19 and ABCB1 genes and individualized treatment with clopidogrel. Pharmacogenomics. 2011 Feb;12(2):141-4. doi: 10.2217/pgs.10.211. No abstract available. PMID 21332306
- [Background] Brandt JT, Close SL, Iturria SJ, Payne CD, Farid NA, Ernest CS 2nd, Lachno DR, Salazar D, Winters KJ. Common polymorphisms of CYP2C19 and CYP2C9 affect the pharmacokinetic and pharmacodynamic response to clopidogrel but not prasugrel. J Thromb Haemost. 2007 Dec;5(12):2429-36. doi: 10.1111/j.1538-7836.2007.02775.x. Epub 2007 Sep 26. PMID 17900275
- [Background] Collet JP, Hulot JS, Pena A, Villard E, Esteve JB, Silvain J, Payot L, Brugier D, Cayla G, Beygui F, Bensimon G, Funck-Brentano C, Montalescot G. Cytochrome P450 2C19 polymorphism in young patients treated with clopidogrel after myocardial infarction: a cohort study. Lancet. 2009 Jan 24;373(9660):309-17. doi: 10.1016/S0140-6736(08)61845-0. Epub 2008 Dec 26. PMID 19108880
- [Background] Mega JL, Close SL, Wiviott SD, Shen L, Hockett RD, Brandt JT, Walker JR, Antman EM, Macias W, Braunwald E, Sabatine MS. Cytochrome p-450 polymorphisms and response to clopidogrel. N Engl J Med. 2009 Jan 22;360(4):354-62. doi: 10.1056/NEJMoa0809171. Epub 2008 Dec 22. PMID 19106084
- [Background] Mega JL, Simon T, Collet JP, Anderson JL, Antman EM, Bliden K, Cannon CP, Danchin N, Giusti B, Gurbel P, Horne BD, Hulot JS, Kastrati A, Montalescot G, Neumann FJ, Shen L, Sibbing D, Steg PG, Trenk D, Wiviott SD, Sabatine MS. Reduced-function CYP2C19 genotype and risk of adverse clinical outcomes among patients treated with clopidogrel predominantly for PCI: a meta-analysis. JAMA. 2010 Oct 27;304(16):1821-30. doi: 10.1001/jama.2010.1543. PMID 20978260
- [Background] Montalescot G, Wiviott SD, Braunwald E, Murphy SA, Gibson CM, McCabe CH, Antman EM; TRITON-TIMI 38 investigators. Prasugrel compared with clopidogrel in patients undergoing percutaneous coronary intervention for ST-elevation myocardial infarction (TRITON-TIMI 38): double-blind, randomised controlled trial. Lancet. 2009 Feb 28;373(9665):723-31. doi: 10.1016/S0140-6736(09)60441-4. PMID 19249633
- [Background] Wallentin L, James S, Storey RF, Armstrong M, Barratt BJ, Horrow J, Husted S, Katus H, Steg PG, Shah SH, Becker RC; PLATO investigators. Effect of CYP2C19 and ABCB1 single nucleotide polymorphisms on outcomes of treatment with ticagrelor versus clopidogrel for acute coronary syndromes: a genetic substudy of the PLATO trial. Lancet. 2010 Oct 16;376(9749):1320-8. doi: 10.1016/S0140-6736(10)61274-3. PMID 20801498
- [Background] Bergmeijer TO, Janssen PW, Schipper JC, Qaderdan K, Ishak M, Ruitenbeek RS, Asselbergs FW, van 't Hof AW, Dewilde WJ, Spano F, Herrman JP, Kelder JC, Postma MJ, de Boer A, Deneer VH, ten Berg JM. CYP2C19 genotype-guided antiplatelet therapy in ST-segment elevation myocardial infarction patients-Rationale and design of the Patient Outcome after primary PCI (POPular) Genetics study. Am Heart J. 2014 Jul;168(1):16-22.e1. doi: 10.1016/j.ahj.2014.03.006. Epub 2014 Mar 21. PMID 24952855
- [Derived] Azzahhafi J, Bergmeijer TO, van den Broek WWA, Chan Pin Yin DRPP, Rayhi S, Peper J, Bor WL, Claassens DMF, van Schaik RHN, Ten Berg JM. Effects of CYP3A4*22 and CYP3A5 on clinical outcome in patients treated with ticagrelor for ST-segment elevation myocardial infarction: POPular Genetics sub-study. Front Pharmacol. 2022 Dec 5;13:1032995. doi: 10.3389/fphar.2022.1032995. eCollection 2022. PMID 36545312
- [Derived] Claassens DMF, van Dorst PWM, Vos GJA, Bergmeijer TO, Hermanides RS, van 't Hof AWJ, van der Harst P, Barbato E, Morisco C, Tjon Joe Gin RM, Asselbergs FW, Mosterd A, Herrman JR, Dewilde WJM, Postma MJ, Deneer VHM, Ten Berg JM, Boersma C. Cost Effectiveness of a CYP2C19 Genotype-Guided Strategy in Patients with Acute Myocardial Infarction: Results from the POPular Genetics Trial. Am J Cardiovasc Drugs. 2022 Mar;22(2):195-206. doi: 10.1007/s40256-021-00496-4. Epub 2021 Sep 7. PMID 34490590
- [Derived] Mahmoodi BK, Eriksson N, Vos GJA, Meijer K, Siegbahn A, James S, Wallentin L, Ten Berg JM. Factor V Leiden Does Not Modify the Phenotype of Acute Coronary Syndrome or the Extent of Myocardial Necrosis. J Am Heart Assoc. 2021 Jun;10(11):e020025. doi: 10.1161/JAHA.120.020025. Epub 2021 May 17. PMID 33998271
- [Derived] Claassens DMF, Bergmeijer TO, Vos GJA, Hermanides RS, van 't Hof AWJ, van der Harst P, Barbato E, Morisco C, Tjon Joe Gin RM, Asselbergs FW, Mosterd A, Herrman JR, Dewilde WJM, Janssen PWA, Kelder JC, Mahmoodi BK, Deneer VHM, Ten Berg JM. Clopidogrel Versus Ticagrelor or Prasugrel After Primary Percutaneous Coronary Intervention According to CYP2C19 Genotype: A POPular Genetics Subanalysis. Circ Cardiovasc Interv. 2021 Apr;14(4):e009434. doi: 10.1161/CIRCINTERVENTIONS.120.009434. Epub 2021 Mar 16. PMID 33722066
- [Derived] Claassens DMF, Vos GJA, Bergmeijer TO, Hermanides RS, van 't Hof AWJ, van der Harst P, Barbato E, Morisco C, Tjon Joe Gin RM, Asselbergs FW, Mosterd A, Herrman JR, Dewilde WJM, Janssen PWA, Kelder JC, Postma MJ, de Boer A, Boersma C, Deneer VHM, Ten Berg JM. A Genotype-Guided Strategy for Oral P2Y12 Inhibitors in Primary PCI. N Engl J Med. 2019 Oct 24;381(17):1621-1631. doi: 10.1056/NEJMoa1907096. Epub 2019 Sep 3. PMID 31479209